CLINICAL TRIAL: NCT01049945
Title: A Phase I/II, Multicenter, Open-label, Dose-escalation Study of Bendamustine in Combination With Lenalidomide and Dexamethasone in Patients With Relapsed Multiple Myeloma
Brief Title: Bendamustine Hydrochloride, Lenalidomide, and Dexamethasone in Treating Patients With Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMRC-020-021; NCI-2009-01535 (Registry Identifier: NCI's CTRO); MMRC-020-021 (Other: Mayo Clinic Cancer Center & MMRC); 09-004211 (Other: Mayo Clinic IRB); C18083/6125 (Other: Cephalon protocol); NCT04567862 (obsolete NCT alias)
Record Dates: First submitted 2010-01-14; First posted 2010-01-15 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2016-04

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bendamustine Hydrochloride; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive dexamethasone orally or IV on days 1, 8, 15, and 22; bendamustine hydrochloride IV over 30 minutes on days 1 and 2; and oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bendamustine hydrochloride; Drug: lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: bendamustine hydrochloride — Given IV
  Other Names: bendamustin hydrochloride; bendamustine; cytostasan hydrochloride; Ribomustin; SDX-105; Treanda
Drug: lenalidomide — Given orally
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: dexamethasone — Given orally or IV
  Other Names: Aeroseb-Dex; Decaderm; Decadron; Decaspray; DM; DXM

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bendamustine hydrochloride and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Lenalidomide may stimulate the immune system in different ways and stop cancer cells from growing. Giving bendamustine hydrochloride together with lenalidomide and dexamethasone may kill more cancer cells. PURPOSE: This phase I/II trial is studying the side effects and best dose of bendamustine hydrochloride and lenalidomide when given together with dexamethasone and to see how well they work in treating patients with relapsed multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the Maximum Tolerated Dose (MTD) of bendamustine and lenalidomide in combination with dexamethasone in subjects with Multiple Myeloma (MM) in first or second relapse. (Phase I) II. To evaluate the confirmed response rate of bendamustine in combination with lenalidomide and dexamethasone in subjects with MM in first or second relapse. (Phase II) SECONDARY OBJECTIVES: I. To evaluate the safety of bendamustine in combination with lenalidomide and dexamethasone. (Phase I and II) II. To evaluate time-to-tumor-progression, progression-free survival, duration of response, and overall survival. (Phase II) OUTLINE: This is a phase I dose escalation study of bendamustine hydrochloride and lenalidomide followed by a phase II study. Patients receive dexamethasone orally or IV on days 1, 8, 15, and 22; bendamustine hydrochloride IV over 30 minutes on days 1 and 2; and oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving at least stable disease after 6 courses may continue to receive lenalidomide and dexamethasone as above in the absence of disease progression or unacceptable toxicity. Dexamethasone may be discontinued after 12 courses of therapy at the treating investigator's discretion. After completion of study treatment, patients are followed at 4 weeks and then periodically for up to 2 years.

ELIGIBILITY:
Inclusion:

* Diagnosis of MM and documentation of at least 1 prior therapy (induction therapy followed by stem cell transplantation is considered one prior therapy) but not more than two previous therapies
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy; all patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information
* Able to take aspirin (325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA or at high risk of developing thrombosis may use warfarin or low molecular weight heparin)
* AST (SGOT) and ALT (SGPT) =< 3.0 x upper limit of normal (ULN)
* Creatinine clearance >= 60 mL/min (Cockcroft-Gault calculation) for patients enrolled in Phase 1 and Creatinine clearance >= 30 mL/min (Cockcroft-Gault calculation) for patients enrolled in phase 2 portion
* Patients with measurable disease, defined by any of the following: serum monoclonal protein >= 1.0 g by protein electrophoresis; > 200 mg of monoclonal protein in the urine on 24-hour electrophoresis; serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio; or monoclonal bone marrow plasmacytosis >= 30% (evaluable disease)
* All necessary baseline studies for determining eligibility must be obtained within 21 days prior to enrollment
* Subject has an ECOG =< 2 OR Karnofsky >= 60% performance status; patients with lower performance status based solely on bone pain secondary to multiple myeloma will be eligible
* FCBP must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing
* Absolute neutrophil count (ANC) >= 1,000 cells/dL (1.0 x 10^9/L) (growth factors cannot be used within 14 days of first drug administration)
* Untransfused platelet count >= 75,000 cells/dL (50 x 10^9/L) for patients in whom < 50% of bone marrow nucleated cells are plasma cells; but platelet count >=50,000/dL for patients in whom 50% of bone marrow nucleated cells are plasma cells
* Total Bilirubin =< 1.5 mg/dL
* Hemoglobin >= 8.0 g/dl

Exclusion:

* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Patients may be receiving concomitant therapy with bisphosphonates and low dose corticosteroids (e.g., prednisone up to but no more than 10 mg p.o. q.d. or its equivalent) for symptom management and comorbid conditions; doses of corticosteroid should be stable for at least 7 days prior to study treatment
* Prior radiation therapy within 2 weeks of the first dose of study treatment
* Known active infection requiring parenteral or oral anti-infective treatment
* Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse follow-up evaluation
* Patient has hypersensitivity to any of the components of study therapy - Known HIV or active hepatitis B or C viral infection
* Known hypersensitivity to required prophylactic medications
* Patient has received other investigational drugs within 14 days before enrollment
* Pregnant or breast-feeding females (lactating females must agree not to breast feed while taking lenalidomide)
* Subjects with evidence of mucosal or internal bleeding and/or platelet transfusion refractory (i.e., unable to maintain a platelet count >= 50,000 cells/mm^3)
* Concurrent therapy with a marketed or investigational anticancer therapy
* Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient
* Other investigational agents are not to be used during the study
* Prior peripheral stem cell transplant within 12 weeks of the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2015-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji K. Kumar, M.D., Study Chair — Mayo Clinic; Vivek Roy, M.D., Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - City of Hope, Duarte, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Washington Universtiy School of Medicine, St Louis, Missouri

REFERENCES:
- [Derived] Kumar SK, Krishnan A, LaPlant B, Laumann K, Roy V, Zimmerman T, Gertz MA, Buadi FK, Stockerl Goldstein K, Birgin A, Fiala M, Duarte L, Maharaj M, Levy J, Vij R. Bendamustine, lenalidomide, and dexamethasone (BRD) is highly effective with durable responses in relapsed multiple myeloma. Am J Hematol. 2015 Dec;90(12):1106-10. doi: 10.1002/ajh.24181. Epub 2015 Oct 6. PMID 26331432

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I, Dose Level 1: Bendamustine 50 mg/m^2 IV day 1 Lenalidomide 15 mg PO days 1-21 Dexamethasone 40 mg PO or IV days 1, 8, 15, 22 Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity
- Phase I, Dose Level 2: Bendamustine 50 mg/m^2 IV day 1 and 2 Lenalidomide 15 mg PO days 1-21 Dexamethasone 40 mg PO or IV days 1, 8, 15, 22 Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity
- Phase I, Dose Level 3: Bendamustine 75 mg/m^2 IV day 1 and 2 Lenalidomide 15 mg PO days 1-21 Dexamethasone 40 mg PO or IV days 1, 8, 15, 22 Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity
- Phase I, Dose Level 4; Phase II, Dose Level 4: Bendamustine 75 mg/m^2 IV day 1 and 2 Lenalidomide 25 mg PO days 1-21 Dexamethasone 40 mg PO or IV days 1, 8, 15, 22 Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity
- Phase I, Dose Level 5: Bendamustine 100 mg/m^2 IV day 1 and 2 Lenalidomide 25 mg PO days 1-21 Dexamethasone 40 mg PO or IV days 1, 8, 15, 22 Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4 | Phase I, Dose Level 5 | Phase II, Dose Level 4
Started | 3 | 6 | 3 | 6 | 3 | 49
Completed | 3 | 6 | 3 | 6 | 3 | 49
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I; Maximum Tolerated Dose, Dose Level 4: Participant demographics were analyzed according to their status for the Phase II Primary Endpoint. All participants registered to Dose Level 4 (the Maximum Tolerated Dose (MTD)) were eligible for the Phase II Primary Endpoint. This group included the 6 patients registered to Phase I, Dose Level 4 and the 49 participants registered to the Phase II portion. The demographic information for all other participants registered to Phase I (Dose Level 1, Dose Level 2, Dose Level 3, and Dose Level 5) were summarized together.
- Total: Total of all reporting groups
Arm/Group | Phase I | Maximum Tolerated Dose, Dose Level 4 | Total
Number analyzed (Participants) | 15 | 55 | 70
Age, Continuous [Median (Full Range); unit: years] | 63.5 [41.8 to 75.0] | 61.9 [40.1 to 86.3] | 62.3 [40.1 to 86.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 27 | 30
  Male | 12 | 28 | 40
Region of Enrollment [Number; unit: participants]
  United States | 15 | 55 | 70

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity of Bendamustine Hydrochloride and Lenalidomide in Combination With Dexamethasone (Phase I)
Description: The Maximum Tolerated Dose (MTD) is the dose level below that at which a dose limiting toxicity (DLT) is observed in ≥ 33% (i.e., ≥ 2 of 6) subjects in a cohort. A dose limiting toxicity is defined as one of the following adverse events in the Common Terminology Criteria for Adverse Events (CTCAE) v 3.0 deemed at least possibly related to treatment:
  * Grade 2 neuropathy with pain
  * Any grade 3 Non-Hematologic toxicity
  * Any grade Non-Hematologic event requiring a dose reduction in cycle 1 or delaying the next cycle by >14 days.
  * Grade 4 neutropenia
  * Febrile neutropenia
  * Grade 4 thrombocytopenia
  * Grade 3 thrombocytopenia associated with bleeding
  * Any Hematologic event requiring a dose reduction in cycle 1 or a delay in the next cycle of treatment by >14 days.
  We are reporting the results of this endpoint as the number of DLTs per dose level.
Time Frame: One cycle of treatment
Population: All participants registered to the Phase I portion of this study were evaluable for this endpoint.
Measure: Number; unit: Dose Limiting Toxic Events
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4 | Phase I, Dose Level 5
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 3
Dose Limiting Toxic Events | 0 | 1 | 0 | 0 | 2

2. Primary Outcome: Confirmed Response Rate (Dose Level 4) Reported as the Percentage of Patients Achieving a Confirmed Response (sCR, CR, VGPR, or PR).
Description: Complete response (CR)
  - Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow.
  Stringent complete response (sCR) - A CR plus normal FLC ratio and no clonal cells in bone marrow
  Near complete response (nCR) A CR, with the persistence of original monoclonal protein
  Very good partial response (VGPR)
  - Serum and urine M-component detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-component plus urine M-component <100 mg per 24 h
  Partial response (PR)
  * ≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200 mg per 24 h.
  * a ≥50% decrease in the difference between involved and uninvolved FLC levels
  * or a ≥50% reduction in plasma cells is required in place of M-protein, if ≥30% at baseline.
Time Frame: Up to 6 cycles of treatment
Population: All participants registered to Dose Level 4 (the Maximum Tolerated Dose (MTD)) were eligible for the Phase II Primary Endpoint. This group included the 6 patients registered to Phase I, Dose Level 4 and the 49 participants registered to the Phase II portion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Maximum Tolerated Dose, Dose Level 4: Bendamustine 75 mg/m^2 IV day 1 and 2 Lenalidomide 25 mg PO days 1-21 Dexamethasone 40 mg PO or IV days 1, 8, 15, 22 Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Maximum Tolerated Dose, Dose Level 4
Number analyzed (Participants) | 55
percentage of participants | 44 [30 to 58]

3. Secondary Outcome: Duration of Response (DOR) (Phase II)
Description: DOR is the time from the date the patient's objective status is first noted to be PR or better to the earliest date of progression (PD=Increase of > 25% from lowest response value in Serum/Urine M-component) is documented. Treatment response was assessed using the International Myeloma Working Group uniform criteria. Complete response (CR)=Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and <5% plasma cells in bone marrow. Stringent complete response (sCR)=A CR plus normal FLC ratio and no clonal cells in bone marrow. Near complete response (nCR)=A CR, with the persistence of original monoclonal protein. Very good partial response (VGPR) =Serum and urine M-component detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-component plus urine M-component <100 mg per 24 h, Partial response (PR)=≥50% reduction of serum M-protein and reduction in 24-h urinary M-protein by ≥90% or to <200 mg per 24 h.
Time Frame: Up to 2 years from study completion
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Maximum Tolerated Dose, Dose Level 4
Number analyzed (Participants) | 55
months | 24.4 [10.8 to 29]

4. Secondary Outcome: Event Free Survival (Phase II)
Description: The event-free survival time is defined as the time from registration to disease progression (PD=Increase of > 25% from lowest response value in Serum/Urine M-component) while receiving bendamustine, lenalidomide, and dexamethasone, death due to any cause, or subsequent treatment for multiple myeloma. The distribution of event-free survival will be estimated using the method of Kaplan-Meier. Treatment response was assessed using the International Myeloma Working Group uniform criteria.
Time Frame: Up to 2 years from study completion
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Maximum Tolerated Dose, Dose Level 4
Number analyzed (Participants) | 55
months | 5.6 [3.2 to 9.1]

5. Secondary Outcome: Progression Free Survival (Phase II)
Description: The progression-free survival time is defined as the time from registration to disease progression (PD=Increase of > 25% from lowest response value in Serum/Urine M-component) while receiving bendamustine, lenalidomide, and dexamethasone or death due to any cause, whichever comes first. The distribution of progression-free survival will be estimated using the method of Kaplan-Meier. Treatment response was assessed using the International Myeloma Working Group uniform criteria.
Time Frame: Up to 2 years from study completion
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Maximum Tolerated Dose, Dose Level 4
Number analyzed (Participants) | 55
months | 11.8 [3.5 to 13.8]

6. Secondary Outcome: Overall Survival (Phase II)
Description: The overall survival time is defined as the time from registration to death due to any cause. The distribution of overall survival will be estimated using the method of Kaplan-Meier. The overall survival rate at 6 months is defined as the percentage of participants who are alive at 6 months.
Time Frame: at 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maximum Tolerated Dose, Dose Level 4
Number analyzed (Participants) | 55
percentage of participants | 87 [77 to 97]

ADVERSE EVENTS:
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4 | Phase I, Dose Level 5 | Phase II, Dose Level 4
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/6 | 2/3 | 2/6 | 1/3 | 24/49
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 6/6 | 3/3 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 (N=3) | Phase I, Dose Level 2 (N=6) | Phase I, Dose Level 3 (N=3) | Phase I, Dose Level 4 (N=6) | Phase I, Dose Level 5 (N=3) | Phase II, Dose Level 4 (N=49)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CNS hemorrhage/bleeding (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I, Dose Level 1 (N=3) | Phase I, Dose Level 2 (N=6) | Phase I, Dose Level 3 (N=3) | Phase I, Dose Level 4 (N=6) | Phase I, Dose Level 5 (N=3) | Phase II, Dose Level 4 (N=49)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (8)
Leg Cramp (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 8 (14)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 22 (25)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Cardiac pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 5 (5)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (5)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 15 (15)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (3) | 1 (1) | 5 (7) | 1 (1) | 24 (26)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 9 (10)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Melena/GI bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 23 (23)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 14 (14)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Edema limbs (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (9)
Fatigue (General disorders) | 3 (4) | 3 (4) | 0 (0) | 4 (4) | 2 (2) | 27 (30)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (11)
Gait abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 4 (5) | 2 (2) | 10 (11)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 11 (12)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (3) | 3 (3) | 3 (3) | 5 (5) | 3 (4) | 39 (39)
Lymphocyte count decreased (Investigations) | 2 (3) | 5 (6) | 3 (3) | 6 (6) | 2 (2) | 42 (43)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 3 (4) | 5 (7) | 3 (4) | 40 (48)
Platelet count decreased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 4 (6) | 1 (1) | 32 (34)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 14 (14)
White blood cell decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 7 (7)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 7 (7)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 10 (11)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 19 (23)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 8 (8)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 8 (8)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (4) | 1 (1) | 14 (14)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 11 (11)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 8 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 10 (11)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes